CLINICAL TRIAL: NCT00983931
Title: A One-Directional, Open-label Drug Interaction Study to Investigate the Effects of Single-Dose Cyclosporine on Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Colchicine and Cyclosporine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1016
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics; Healthy
Keywords: healthy; adult; colchicine; cyclosporine; blood levels over time
MeSH Terms: interventions — Colchicine; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): -baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Cyclosporine (Experimental): -colchicine pharmacokinetics in presence of cyclosporine
  Interventions: Drug: Cyclosporine; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone at 7:15 a.m. on Day 1 after an overnight fast of at least 10 hours.
  Other Names: COLCRYS™
  Arms: Colchicine alone
Drug: Cyclosporine — A single dose of 100 mg cyclosporine administered with colchicine at 7:15 a.m. on Day 15 after an overnight fast of at least 10 hours.
  Other Names: Neoral® (Novartis Pharmaceuticals Corporation)
  Arms: Colchicine with Cyclosporine
Drug: Colchicine — A single dose of 0.6 mg colchicine administered with cyclosporine at 7:15 a.m. on Day 15 after an overnight fast of at least 10 hours.
  Arms: Colchicine with Cyclosporine

SUMMARY:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Cyclosporine is a potent inhibitor of both CYP3A4 and P-gp. This study will evaluate the effect of single-dose cyclosporine on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period

DETAILED DESCRIPTION:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Cyclosporine is a potent inhibitor of both CYP3A4 and P-gp. This study will evaluate the effect of single-dose cyclosporine on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. On study Day 1 after a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of colchicine (1 x 0.6 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis on Days 2-5. A 14 day washout period will be completed after the first dose of colchicine on Day 1. On Day 15 after a fast of at least 10 hours, all study participants will receive co-administered single oral doses of colchicine (1 x 0.6 mg tablet) and cyclosporine (1 x 100 mg capsule). Fasting will continue for 4 hours after the dose. Subjects will be confined to the clinic for dosing and a 24 hour period after the dose. Blood samples will be drawn from all participants before dosing and during the 24 hour post-dose period at times sufficient to adequately determine the pharmacokinetics of colchicine. Blood sampling will continue on a non-confined basis on Days 16-19. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (blood pressure and pulse) will be measured prior to dosing and at 1, 2, and 3 hours following drug administration on Days 1 and 15 to coincide with peak plasma concentrations of both colchicine and cyclosporine. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive.

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine or cyclosporine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R G, Pharm.D., Principal Investigator — PRACS - Cetero
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Wason S, Digiacinto JL, Davis MW. Effect of cyclosporine on the pharmacokinetics of colchicine in healthy subjects. Postgrad Med. 2012 Jul;124(4):189-96. doi: 10.3810/pgm.2012.07.2579. PMID 22913907
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, male and female volunteers, consisting of volunteers from the community at large, were enrolled in the study.
Pre-assignment Details: 41 subjects were screened, 11 were screen failures, 4 had schedule conflicts, 1 was transferred to a different study, and 1 was not needed
Groups:
- Colchicine Alone / With Cyclosporine: [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days. Then, on Day 15, each subject received both one 0.6 mg colchicine tablet and one 100 mg cyclosporine capsule at 7:15 a.m. after an overnight fast of at least 10 hours.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Cyclosporine
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Cyclosporine
Started | 24
Completed | 23 (one subject withdrawn due to creatine kinase out of range)
Not Completed | 1
Not completed — Physician Decision | 1
Period: Colchicine With Cyclosporine
Arm/Group | Colchicine Alone / With Cyclosporine
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone / With Cyclosporine
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] — age range: >=18 and <=45 years old
  years | 29.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to colchicine dosing on Days 1 and 15, and then 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours after colchicine dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:15 a.m. after an overnight fast, followed by a washout period of 14 days.
- Colchicine With Cyclosporine: On Day 15, each subject received both one 0.6 mg colchicine tablet and one 100 mg cyclosporine capsule at 7:15 a.m. after an overnight fast of at least 10 hours.
Arm/Group | Colchicine Alone | Colchicine With Cyclosporine
Number analyzed (Participants) | 23 | 23
pg/mL | 2,720.04 (1,137.85) | 8,817.48 (2,223.80)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Cyclosporine
Number analyzed (Participants) | 23 | 23
pg-hr/mL | 12,545.04 (5,854.46) | 39,828.11 (10,312.85)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Cyclosporine
Number analyzed (Participants) | 23 | 23
pg-hr/mL | 14,996.79 (7,789.77) | 47,312.02 (12,137.79)

ADVERSE EVENTS:
Arm/Group | Colchicine Alone | Colchicine With Cyclosporine
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 4 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Colchicine With Cyclosporine
abdominal pain upper (Gastrointestinal disorders) | 0/24 (0) | 1/23 (1)
nausea (Gastrointestinal disorders) | 1/24 (1) | 0/23 (0)
bacteriuria (Infections and infestations) | 1/24 (1) | 0/23 (0)
contusion (Injury, poisoning and procedural complications) | 1/24 (1) | 0/23 (0)
dizziness (Nervous system disorders) | 1/24 (1) | 0/23 (0)
headache (Nervous system disorders) | 1/24 (1) | 3/23 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/23 (1)
pharynolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/24 (1) | 0/23 (0)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 0/24 (0) | 1/23 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days